CLINICAL TRIAL: NCT00506532
Title: The Use of Surfactant in Lung Transplantation: A Randomized Control Pilot Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMC063344ctil
Record Dates: First submitted 2007-07-15; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Lung Transplantation; Primary Graft Dysfunction
Keywords: Pulmonary Surfactants; Lung transplantation; Primary Graft Dysfunction
MeSH Terms: conditions — Primary Graft Dysfunction | interventions — Surface-Active Agents; calfactant

INTERVENTIONS:
Drug: Surfactant (calfactant)

SUMMARY:
1. Working Hypothesis:

   The purpose of the trial is to study the effect of exogenous calf surfactant (calfactant) on the prevention of primary graft failure due to ischemic-reperfusion lung injury in lung transplant patients.
2. Aims of the Study:

The purpose of the trial is to study the effect of exogenous calf surfactant (calfactant) on the prevention of primary graft failure due to ischemic-reperfusion lung injury in lung transplant patients.

DETAILED DESCRIPTION:
Background: Lung transplantation induces surfactant dysfunction that may be a contributing factor for primary graft dysfunction (PGD) and graft failure. Animal studies and limited human reports suggest that surfactant administration may prevent primary graft dysfunction.

Working hypothesis and aims:

The purpose of the trial is to study the effect of exogenous calf surfactant (calfactant) on the prevention of primary graft failure due to ischemic-reperfusion lung injury in lung transplant patients.

Methods: The trial is an open randomized controlled prospective study. Patient population: 42 patients eligible for lung transplant according to hospital criteria.

Study medication: Calfactant intratracheal suspension -an extract of natural surfactant from calf lungs, which includes phospholipids, neutral lipids and surfactant-associated proteins B and C (SP-B and SP-C).

Study design: Patients randomized to receive calfactant will have the drug administered through a fiberoptic bronchoscope distributing the drug evenly across the lung immediately after connection. The other patient will not have any administration to avoid any excessive flushing. When 2 lungs will be used from the same donor for 2 recipients one patient receiving one lung will be treated with calfactant while the other patient receiving the other lung will not be treated and serve as the control. Otherwise lungs will be treated with surfactant in every other case.

Expected results: We expect surfactant instillation during lung transplantation to improve oxygenation, prevent primary graft dysfunction, make intubation time shorter and to enhance early post transplantation recovery. In a pilot study that we already performed results are encouraging.

Importance: PGD could cause substantial morbidity and mortality among transplanted patients. In a pilot study we already found that surfactant instillation during lung transplantation improves oxygenation, prevents primary graft dysfunction, shortens intubation time and ICU stay. We believe that surfactant treatment enhances early post transplantation recovery, and may also be cost effective by shortening expensive ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for lung transplantation

Exclusion Criteria:

* Differential diagnosis of PGD
* Pulmonary Edema
* Stenosis or thrombosis of pulmonary artery/vein anastomosis

Ages: 16 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Effect of intraoperative exogenous surfactant treatment on oxygenation and primary graft dysfunction (PGD) prevention (primary outcome) | 3 days post operation

SECONDARY OUTCOMES:
Recovery-Extubation ;Seating time; Icu stay; Hospital stay; Lung function | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: MordechaI R Kramer, Prof, Principal Investigator — Pulmonary Institute Rabin Medical Center
Locations (1):
- Pulmonary Institute Rabin Medical Center, Petah Tikva, Israel